CLINICAL TRIAL: NCT04652375
Title: Outcomes After Albumin Vs Lactated Ringer's Solution in CABG and AVR Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2000025462; 000 (Other: 11.8.23)
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Bypass Graft Surgery; Aortic Valve Replacement
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albumin Solution (Experimental): Participants will receive Albumin solution for fluid resuscitation post-surgery.
  Interventions: Other: Albumin Solution
- Lactated Ringer's Solution (Experimental): Participants will receive lactated Ringer's for fluid resuscitation post-surgery
  Interventions: Other: Lactated Ringer's Solution

INTERVENTIONS:
Other: Albumin Solution — Participants will receive Albumin solution for fluid resuscitation post-surgery.
  Arms: Albumin Solution
Other: Lactated Ringer's Solution — Participants will receive Lactated Ringer's solution for fluid resuscitation post-surgery.
  Arms: Lactated Ringer's Solution

SUMMARY:
This is a prospective, randomized, double-blinded study to compare the use of albumin versus lactated Ringer's solution in patients undergoing coronary artery bypass graft surgery and in patients undergoing aortic valve replacement surgery and evaluate the incidence of acute kidney injury as a primary outcome.

DETAILED DESCRIPTION:
This will be a prospective, randomized, double-blinded study to compare the use of albumin versus lactated Ringer's solution in patients undergoing coronary artery bypass graft surgery and in patients undergoing aortic valve replacement surgery and evaluate the incidence of acute kidney injury as a primary outcome. Data will be collected from both EPIC and STS (society of thoracic surgeons) database. STS database extracts data from the electronic medical record and groups it in specific format to evaluate outcomes after cardiac surgery to compare institutional performance to similar institutions and the national average. Patients undergoing coronary artery bypass graft or aortic valve replacement will be randomized to receive either albumin or lactated Ringer's for fluid resuscitation post-surgery. The resuscitation volume will be based on clinical decision after examining all the hemodynamics parameters. This practice coincides with standard of care and current practice. All eligible patients will be randomly assigned to receive either albumin 5% or lactated Ringer's solution in a 1:1 ratio using computer-generated, permutated blocks of 2 - 4. Both solutions will be administered intravenously in 250 mL increments at the discretion of the physician until hemodynamic parameters are met. The IV infusion bag and IV tubing will be covered using opaque bags to allow for blinding.

ELIGIBILITY:
Inclusion Criteria:

* All patients greater than 18 years of age undergoing CABG and AVR procedures

Exclusion Criteria:

* Low ejection fraction (<20%) End stage renal disease Chronic renal insufficiency Pre-operative Inotropic (eg. Dobutamine) or vasoactive IV infusions (e.g, norepinephrine)

  * Jehovah's Witness Emergent surgery (e.g, intra-aortic balloon pump) Pre-operative acute kidney injury based on AKIN criteria Non English speaking patients
  * Jehovah's Witness population will be excluded regardless of their preference with accepting Albumin because sometimes PRBC are used as part of ongoing resuscitation in bleeding patients and if patients cannot use blood, this will have a much bigger issue with resuscitation and this study is not designed to follow up that population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | Within 72 hours post randomization
  Acute kidney injury will be assessed by these criteria: Stage I. Increase 1.5-1.9 times from baseline or ≥ 0.3 mg/dl increase within 48 h. Urinary output (UOP) < 0.5 ml/kg/h for 6-12 hours Stage II. Increase > 2- to 3-fold from baseline. UOP < 0.5 ml/kg/h for 12 hours Stage III. Increased > 300% (> 3-fold) from baseline, or ≥ 4.0 mg/dl with an acute increase of ≥ 0.5 mg/dl or on renal replacement therapy. UOP < 0.3 ml/kg/h for 24 hours or anuria for 12 hours

SECONDARY OUTCOMES:
Extubation time | Up to 90 days
  Duration of intubation
Length of stay in the ICU | Up to 90 days
  Length of stay in the ICU
Length of stay in the hospital | Up to 90 days
  Length of stay in the hospital
Hospital readmission | Readmission within 30 days of discharge
  An episode when a patient who had been discharged from a hospital is admitted again within a specified time interval

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Tantway, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No